CLINICAL TRIAL: NCT06349265
Title: A Comparative Analysis of the Efficacy of Ultrasound-Guided Injection of 5% Dextrose in Water for the Treatment of Mild to Severe Carpal Tunnel Syndrome
Brief Title: Ultrasound-Guided 5% Dextrose Injection for Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Gamze Gul Gulec, Assistant Proffesor, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Carpal Tunnel Syndrome
Keywords: dextrose; carpal tunnel syndrome; ultrasound
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Water

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Mild Carpal Tunnel syndrome
  Interventions: Drug: Carpal Tunnel Hydrodissection with %5 dextrose in water injection
- Group 2 (Active Comparator): Moderate Carpal Tunnel Syndrome
  Interventions: Drug: Carpal Tunnel Hydrodissection with %5 dextrose in water injection
- Group 3 (Active Comparator): Severe Carpal Tunnel Syndrome
  Interventions: Drug: Carpal Tunnel Hydrodissection with %5 dextrose in water injection

INTERVENTIONS:
Drug: Carpal Tunnel Hydrodissection with %5 dextrose in water injection — Under the inplane ulnar approach, 3ml injectate was injected to hydrodissect the median nerve from the flexor retinaculum, and the residual 2ml injectate was then injected to hydrodissect the inferior median nerve away from the flexor tendons.

SUMMARY:
This study was a prospective randomized double-blind clinical trial conducted at the Physical Medicine and Rehabilitation Clinic of a local research and training hospital in Turkey from October 2023 and May 2024. Patients diagnosed with CTS were classified into three groups: severe, mild, and moderate CTS, based on the results of electrophysiological tests. An ultrasound-guided 5% Dextrose in Water injection was performed. The primary outcome measurement was the Visual Analog Scale (VAS), while secondary measurements were the Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) and the Dolour Neuropathic en 4 Questions (DN4) questionnaire. The measurements were performed before the injection and at the first week, first month and third month follow-up times. The distribution of data within groups was examined using the Shapiro-Wilk test and Q-Q plots. The study also analyzed temporal changes, group differences, and intergroup changes using repeated measures ANOVA models.

ELIGIBILITY:
Inclusion Criteria:

1. Paresthesia/dysesthesia, painful swelling with clumsy weakness of the hand exacerbated by sleep or repetitive use of the wrist, and relieved by shaking the hand with postural change.
2. Sensory loss with numbness in the median nerve-innervated regions of the hand.
3. Weakness with atrophy of the median nerve-innervated thenar muscles.
4. Positive Phalen's test and/or Tinel's sign.
5. The diagnosis should be confirmed with electrodiagnostic studies.

Exclusion Criteria:

1. History of cervical myelomalacia, polyneuropathy, brachial plexopathy, or thoracic outlet syndrome.
2. History of systematic infection, and rheumatologic disorders.
3. Previous steroid injection for carpal tunnel syndrome.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-03-02 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale(VAS) | At the beginning, 1.,4., 12. week
  VAS is comprised of a horizontal line of 10 cm in length. A measurement of 0 cm indicates the absence of pain, whereas a measurement of 10 cm signifies the most severe pain that one can conceive. Patients are instructed to assess the intensity of discomfort by indicating a point on this line. The Turkish version of the assessment has been validated and shown to be reliable.

SECONDARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) | At the beginning, 1.,4., 12. week
  The Boston Carpal Tunnel Questionnaire (BCTQ) comprises two subscales. The Symptom Severity Scale provides data on symptom intensity, while the Functional Status Scale assesses hand function. The Symptom Severity Scale comprises 11 items evaluating pain, paresthesia, numbness, weakness, night symptoms, and difficulty grasping. Meanwhile, the Functional Status Scale includes eight items assessing functional deficits in writing, buttoning clothes, holding a book while reading, gripping a phone handle, opening jars, performing household chores, carrying a shopping bag, bathing, and dressing.
  Each item is scored from 1 (no symptoms/no difficulty) to 5 (worst symptom or cannot perform the activity at all). The average score of each scale yields a score between 1 and 5, with higher scores indicating more severe symptoms or functional impairments.A Turkish validity and reliability study has been conducted.
Dolour Neuropathique en 4 Questions (DN4) questionnaire | At the beginning, 1.,4., 12. week
  The DN4 (Dolour Neuropathique en 4 Questions) questionnaire is a screening tool designed to aid in diagnosing neuropathic pain. Developed in 2005, it consists of ten items, with seven questions focusing on sensory symptoms and three on signs related to neuropathic pain. The questions cover various characteristics of neuropathic pain, such as burning, tingling, and sensitivity to touch. Turkish validity and reliability measures were established for its use.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Özmen, Study Chair — İstanbul Physical Medicine and Rehabilitation Hospital
Locations (1):
- Gamze Gül Güleç, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No